CLINICAL TRIAL: NCT04603326
Title: FoxBioNet: ECV (Extracellular Vesicle) 004
Status: Completed | Type: Observational
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Collaborators: Indiana University (Other); University of Rochester (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Connie Marras, Associate Professor at University Health Network, University of Toronto, University Health Network, Toronto
Other Study IDs: ECV-004
Record Dates: First submitted 2020-10-23; First posted 2020-10-26 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Biomarker; LRRK2; CSF
MeSH Terms: conditions — Parkinson Disease | interventions — Spinal Puncture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cerebro-Spinal Fluids Immune Cell Collection from Whole Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Non-manifesting LRRK2 mutation carriers: Patients must have confirmed LRRK2 G2019S mutation Age 30 years or older at date of informed consent.
  Interventions: Procedure: Lumbar Puncture
- LRRK2 Parkinson Disease (PD) Participants:: Patients must have confirmed LRRK2 G2019S mutation Patients must meet the MDS criteria for Parkinson's disease Disease duration: any Age 30 years or older at time of PD diagnosis.
  Interventions: Procedure: Lumbar Puncture
- Idiopathic PD (iPD) Particpants:: Patients must meet the MDS criteria for Parkinson's disease. Disease duration: any Age 30 years or older at time of PD diagnosis.
  Interventions: Procedure: Lumbar Puncture
- Control (C) Participants:: Age 30 years or older at date of informed consent.
  Interventions: Procedure: Lumbar Puncture

INTERVENTIONS:
Procedure: Lumbar Puncture — Lumbar Puncture for collection of Cerebrospinal Fluids
  Other Names: Whole Blood Collection

SUMMARY:
The goal of this study is to identify reliable markers of LRRK2 activity in human CSF.

DETAILED DESCRIPTION:
Specific aims of this project are:

Primary Objectives:

To evaluate each assay performance for its ability to detect LRRK2, its activity and/or the detection and activity of the pathways it impacts using a variety of different approaches (quantitative western blot, immunoassays and LC-MS). Assay performance will be assessed and those demonstrating high sensitivity and consistency will be considered for further development.

Secondary Objectives:

To assess the ability of the assay or a combination of assays to differentiate pathogenic LRRK2 variant manifesting and non-manifesting carriers, idiopathic PD and healthy non-carriers.

ELIGIBILITY:
Non-manifesting LRRK2 mutation carriers

Inclusion:

* Ability to provide informed consent
* Confirmed LRRK2 G2019S mutation
* Age 30 years or older at date of informed consent.

Exclusion:

* Inability to provide informed consent
* Known GBA mutation carrier
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans. Participants that have had a 6 - month washout period between ending participation in a clinical trial with an investigational agent and enrollment into the ECV-004 study are eligible.
* The presence of rest tremor, bradykinesia or rigidity.
* The presence of any other neurological sign that in the opinion of the site investigator raises suspicion for an atypical parkinsonian syndrome (e.g. supranuclear gaze palsy)
* Treatment for cancer in the last 5 years or cancer patient receiving immunotherapy or targeted therapy. Individuals with cancers that have not been treated with systemic chemotherapy, immunotherapy, targeted therapies or radiation therapy are eligible to enroll in the study.
* Diagnosis of an autoimmune disorder
* Current treatment with anticoagulants that might preclude safe completion of the lumbar puncture and that cannot be safely paused in the opinion of the site investigator.
* Any condition that, in the investigator's opinion, precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Diagnosis of dementia
* Pregnant females, if fluoroscopy is needed to obtain the spinal fluid sample

LRRK2 Parkinson Disease (PD) Participants:

Inclusion:

* Ability to provide informed consent
* Confirmed LRRK2 G2019S mutation
* Meet the MDS criteria for Parkinson's disease
* Disease duration: any
* Age 30 years or older at time of PD diagnosis.

Exclusion:

* Known GBA mutation carrier
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans. Participants that have had a 6 - month washout period between ending participation in a clinical trial with an investigational agent and enrollment into the ECV-004 study are eligible.
* Treatment for cancer in the last 5 years or cancer patient receiving immunotherapy or targeted therapy. Individuals with cancers that have not been treated with systemic chemotherapy, immunotherapy, targeted therapies or radiation therapy are eligible to enroll in the study.
* Diagnosis of an autoimmune disorder
* Current treatment with anticoagulants that might preclude safe completion of the lumbar puncture and that cannot be safely paused in the opinion of the site investigator.
* Any condition that, in the investigator's opinion, precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Diagnosis of dementia
* Pregnant females, if fluoroscopy is needed to obtain the spinal fluid sample

Idiopathic PD (iPD) Particpants:

Inclusion:

* Ability to provide informed consent
* Meet the MDS criteria for Parkinson's disease.
* Disease duration: any
* Age 30 years or older at time of PD diagnosis.

Exclusion:

* Known LRRK2 G2019S and/or GBA mutation carrier
* Participation in a blinded clinical trial of any kind or an unblinded trial of an investigational product that is not currently approved for use in humans. Participants that have had a 6 - month washout period between ending participation in a clinical trial with an investigational agent and enrollment into the ECV-004 study are eligible.
* Treatment for cancer in the last 5 years or cancer patient receiving immunotherapy or targeted therapy. Individuals with cancers that have not been treated with systemic chemotherapy, immunotherapy, targeted therapies or radiation therapy are eligible to enroll in the study.
* Diagnosis of an autoimmune disorder
* Current treatment with anticoagulants that might preclude safe completion of the lumbar puncture and that cannot be safely paused in the opinion of the site investigator.
* Any condition that, in the investigator's opinion, precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Diagnosis of dementia
* Pregnant females, if fluoroscopy is needed to obtain the spinal fluid sample

Control (C) Participants:

Inclusion:

* Ability to provide informed consent
* Age 30 years or older at date of informed consent.

Exclusion:

* Known GBA mutation carrier
* In the absence of prior genetic testing for LRRK2 G2019S mutations: Family history of Parkinson's disease is an exclusion criterion. If genetic testing for LRRK2 G2019S mutations has been performed and is negative, individuals with a family history of PD may be enrolled.
* The presence of rest tremor, bradykinesia or rigidity.
* The presence of any other neurological sign that in the opinion of the site investigator raises suspicion for an atypical parkinsonian syndrome (e.g. supranuclear gaze palsy)
* Treatment for cancer in the last 5 years or cancer patient receiving immunotherapy or targeted therapy. Individuals with cancers that have not been treated with systemic chemotherapy, immunotherapy, targeted therapies or radiation therapy are eligible to enroll in the study.
* Diagnosis of an autoimmune disorder.
* Current treatment with anticoagulants that might preclude safe completion of the lumbar puncture and that cannot be safely paused in the opinion of the site investigator.
* Any condition that, in the investigator's opinion, precludes the safe performance of routine lumbar puncture, such as prohibitive lumbar spinal disease, bleeding diathesis, or clinically significant coagulopathy or thrombocytopenia.
* Diagnosis of dementia
* Pregnant females, if fluoroscopy is needed to obtain the spinal fluid sample

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Approximately 140 participants will be enrolled to participate in this study, with a goal of enrolling 30 non-manifesting LRRK2 carriers, 30 LRRK2 Parkinson's Disease (PD), 40 idiopathic PD, and 40 healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Assay Evaluation | 1 year
  Evaluate each assay performance for ability to detect LRRK2, its activity and/or the detection and activity of the pathways it impacts using a variety of different approaches (quantitative western blot, immunoassays and LC-MS).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Northwestern University, Chicago, Illinois
  - The Trustees of Columbia University, New York, New York
  - Oregon Health Sciences Univeristy, Portland, Oregon
  - The Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania